CLINICAL TRIAL: NCT00173030
Title: Genetic Study of Atrial Fibrillation: Focusing on Renin-Angiotensin System and C-Reactive Protein Genes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700499
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Multi-locus and multi-gene studies of atrial fibrillation, focusing on renin-angiotensin system genes and C reactive protein gene

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation

Exclusion Criteria:

* Patients with atrial fibrillation who are reluctant for the study

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jiunn-Lee Lin, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan